CLINICAL TRIAL: NCT03515876
Title: The Effects of Dexmedetomidine on Segmental EEG Power Spectra Activity Under Propofol-based Anesthesia
Brief Title: Dexmedetomidine on Segmental EEG Power Spectra
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhiyi Zuo (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Zhiyi Zuo, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2018-52
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia; EEG Power Spectra

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients will receive intravenous propofol infusion.
- Dexmedetomidine 0.5 microgram/kg group: Patients will receive dexmedetomidine 0.5 microgram/kg and then intravenous propofol infusion.
- Dexmedetomidine 1 microgram/kg group: Patients will receive dexmedetomidine 1 microgram/kg and then intravenous propofol infusion.

SUMMARY:
To compare the EEG power spectra activity during propofol-based anesthesia in the presence or absence of dexmedetomidine in patients undergoing hysteroscopic examination and surgery to determine whether the addition of dexmedetomidine will induce better sleep-like anesthesia status.

DETAILED DESCRIPTION:
Three groups of patients undergoing hysteroscopic examination and surgery will be studied: 1) control group, patients will receive propofol intravenous infusion to provide anesthesia; 2) dexmedetomidine 0.5 microgram/kg group. This dexmedetomidine dose is infused within 10 min and then the use of propofol for anesthesia; and 3) dexmedetomidine 1 microgram/kg group. This dexmedetomidine dose is infused within 10 min and then the use of propofol for anesthesia.

Each group will have 20 patients.

General conditions including blood pressure, respiration, and heart rates will be recorded.

EEG power spectra activity will be recorded no-invasively by a Narcotrend EEG monitor.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical status I to II grade.
* body mass index 18 to 25 kg/m2
* no vision or hearing impairment
* will receive general anesthesia

Exclusion Criteria:

* with psychological or mental diseases
* with neurological diseases
* treating with steroids or with alcohol dependence.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients undergoing hysteroscopic examination and surgery.
Study Population: patients for hysteroscopic examination and surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
EEG power spectra | From prior to anesthesia to 10 min after anesthesia.
  EEG power spectra monitored no-invasively by Narcotrend

SECONDARY OUTCOMES:
Blood pressure | From prior to anesthesia to 10 min after anesthesia.
  Blood pressure monitored no-invasively
Respiration | From prior to anesthesia to 10 min after anesthesia.
  Monitored no-invasively
Heart rates | From prior to anesthesia to 10 min after anesthesia.
  Monitored no-invasively

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China